CLINICAL TRIAL: NCT04680442
Title: Safety of Continuing HER-2 Directed Therapy in Overt Left Ventricular Dysfunction: A Randomized, Controlled Trial
Brief Title: Safety of Continuing HER-2 Directed Therapy in Overt Left Ventricular Dysfunction
Acronym: SCHOLAR-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRI.SCHOLAR-2
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Heart Failure
MeSH Terms: conditions — Breast Neoplasms; Heart Failure | interventions — Trastuzumab; Ogivri; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Recommendations for continuing or holding trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) for the control group are guided by an adaptation of the 2008 Canadian recommendations.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Trastuzumab emtansine
- Intervention Group (Experimental): The intervention group will continue to receive trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) in the setting of asymptomatic decline in LVEF up to an LVEF of 40% as outlined in the criteria listed in Table 3. For reasons of practicality, in the intervention group, the first dose of trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) after randomization can be administered up to 3 weeks late. This will allow time for the participant to be reviewed by a cardiologist and to receive ACE-I/angiotensin receptor blocker and/or beta-blocker, and for dose titration.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab is a HER-2 targeting monoclonal antibody that improves overall survival and reduces the risk of recurrent disease in early stage HER-2 positive breast cancer.
  Other Names: Herceptin, Herzuma, Ogivri, Trazimera, Kanjinti
Drug: Pertuzumab — Pertuzumab (also called 2C4, trade name Perjeta) is a monoclonal antibody used in combination with trastuzumab and docetaxel for the treatment of metastatic HER2-positive breast cancer; it also used in the same combination as a neoadjuvant in early HER2-positive breast cancer
  Other Names: Perjeta
Drug: Trastuzumab emtansine — Ado-trastuzumab emtansine is approved to treat: Breast cancer that is HER2 positive and has already been treated with a taxane and trastuzumab.
  Other Names: Kadcyla,

SUMMARY:
Trastuzumab is an important treatment for HER 2 positive breast cancer. But trastuzumab can cause injury to the heart, and this is one of the main reasons it cannot be administered as planned. Heart injury can often be successfully treated using cardiac medications. The objectives of SCHOLAR-2 are to evaluate whether is it safe and effective to continue trastuzumab, pertuzumab or trastuzumab-emtansine (T-DM1) in patients with early stage HER-2 positive breast cancer despite mild, minimally symptomatic or asymptomatic systolic left ventricular dysfunction as compared with a guideline-driven approach of withholding or discontinuing trastuzumab, pertuzumab or trastuzumab-emtansine (T-DM1).

In SCHOLAR-2, we will compare two thresholds of withholding or discontinuing trastuzumab/pertuzumab/trastuzumab-emtansine: a threshold that is currently advocated for by existing treatment practice guidelines versus a more aggressive threshold that allows trastuzumab/pertuzumab/trastuzumab-emtansine to continue at lower levels of LVEF than currently supported by guideline documents.

DETAILED DESCRIPTION:
SCHOLAR-2 is a Phase II open-label randomized controlled trial with blinded outcome event ascertainment with a target sample size of 130.

Control Group Recommendations for continuing or holding trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) for the control group are guided by an adaptation of the 2008 Canadian recommendations.

Intervention Group The intervention group will continue to receive trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) in the setting of asymptomatic decline in LVEF up to an LVEF of 40% as outlined in the criteria listed in Table 3. For reasons of practicality, in the intervention group, the first dose of trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) after randomization can be administered up to 3 weeks late. This will allow time for the participant to be reviewed by a cardiologist and to receive ACE-I/angiotensin receptor blocker and/or beta-blocker, and for dose titration.

Study assessments will occur:

1. 3 weeks after randomization
2. 6 weeks after randomization
3. Follow-up at every 3 months thereafter until 12 months after the last dose of trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1)

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-III HER-2 positive breast cancer
2. Receiving adjuvant or neoadjuvant therapy with trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1)
3. Evidence of left ventricular dysfunction, as defined by at least one of:

   a) LVEF < 54% or b) LVEF ≥54% and either i) fall in LVEF of ≥15% from prior to trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) exposure, or ii) New York Heart Association (NYHA) class II heart failure symptoms within the past 6 months

Exclusion Criteria:

1. Current use of both angiotensin converting enzyme inhibitor (ACEI) /angiotensin receptor blocker (ARB) and beta-blocker
2. Contra-indication to both ACE-I/ARB and beta-blockers
3. NYHA class III or IV heart failure
4. LVEF <40%
5. Systolic blood pressure <100mmHg
6. Current or planned pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
primary efficacy outcome | one year
  the proportion of participants completing trastuzumab, pertuzumab, or trastuzumab-emtansine (T-DM1) as planned at its initiation
co-primary safety outcomes | one year
  1. LVEF at the close-out visit, and
  2. The composite of NYHA class III or IV heart failure or cardiovascular death.

SECONDARY OUTCOMES:
secondary outcome measures the composite of NYHA class III or IV heart failure, breast cancer relapse, or all-cause mortality. | one year
  the composite of NYHA class III or IV heart failure, breast cancer relapse, or all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Leong, PhD. MBBSm, Principal Investigator — McMaster University; Som Mukherjee, MD MSc FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (8):
- Brazil (4):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade Da Santa Casa De Misericórdia De Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Clínica de Pesquisa e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo, São Paulo
- Canada (3):
  - Juravnski Cancer Centre, Hamitlon, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
- E.Meshalkin National medical research center of the Ministry of Health of the Russian Federation, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No